Official Title: Revolutionizing Normative Re-education: Delivering Enhanced PNF Within a Social Media Inspired Game About College Life

Document Date: March 1, 2020

## **Consent Forms**

## CampusGANDR App TERMS OF SERVICE & PRIVACY POLICY

- Basic consent for app use and competition participation.
- Format and language consistent IOS and Android app store requirements

INFORMED CONSENT FORM FOR THE EVALUATION STUDY (RCT)

# CAMPUSGANDR TERMS OF SERVICE & PRIVACY POLICY

BY CREATING A CAMPUSGANDR ACCOUNT, THESE TERMS WILL AUTOMATICALLY APPLY TO YOU – YOU SHOULD MAKE SURE THEREFORE THAT YOU READ THEM CAREFULLY BEFORE CREATING AN ACCOUNT. WE ARE OFFERING YOU THIS APP TO USE FOR YOUR OWN PERSONAL USE WITHOUT COST, BUT YOU SHOULD BE AWARE THAT YOU'RE NOT ALLOWED TO COPY, OR MODIFY THE APP, ANY PART OF THE APP, OR OUR TRADEMARKS IN ANY WAY. YOU'RE NOT ALLOWED TO ATTEMPT TO EXTRACT THE SOURCE CODE OF THE APP, AND YOU ALSO SHOULDN'T TRY TO TRANSLATE THE APP INTO OTHER LANGUAGES, OR MAKE DERIVATIVE VERSIONS. THE APP ITSELF, AND ALL THE TRADE MARKS, COPYRIGHT, DATABASE RIGHTS AND OTHER INTELLECTUAL PROPERTY RIGHTS RELATED TO IT. STILL BELONG TO THE CAMPUSGANDR TEAM.

THE CAMPUSGANDR APP STORES AND PROCESSES PERSONAL DATA THAT YOU HAVE PROVIDED TO US SO THAT YOU CAN TAKE PART IN A COMPETITION AT YOUR UNIVERSITY. ACCEPTABLE USE OF THE CAMPUSGANDR APPLICATION, AS WELL AS RULES AND REGULATIONS REGARDING COMPETITIONS AT SPECIFIC UNIVERSITIES ARE DETAILED BELOW. DATA COLLECTED AND STORED BY THE APP ARE DETAILED IN THE PRIVACY POLICY THAT FOLLOWS. IT'S YOUR RESPONSIBILITY TO KEEP YOUR PHONE AND ACCESS TO THE APP SECURE. WE THEREFORE RECOMMEND THAT YOU DO NOT JAILBREAK OR ROOT YOUR PHONE, WHICH IS THE PROCESS OF REMOVING SOFTWARE RESTRICTIONS AND LIMITATIONS IMPOSED BY THE OFFICIAL OPERATING SYSTEM OF YOUR DEVICE. IT COULD MAKE YOUR PHONE VULNERABLE TO MALWARE/VIRUSES/MALICIOUS PROGRAMS, COMPROMISE YOUR PHONE'S SECURITY FEATURES AND IT COULD MEAN THAT THE CAMPUSGAND APP WON'T WORK PROPERLY OR AT ALL.

## **ACCEPTABLE USE**

CAMPUSGANDR OFFERS A FUN WAY FOR NEW COLLEGE STUDENTS TO LEARN ABOUT FELLOW STUDENTS AT THEIR SCHOOL AND LIFE ON THEIR CAMPUS WHILE TESTING THEIR SOCIAL PERCEPTIONS AND COMPETING FOR CASH PRIZES. TO USE CAMPUSGANDR YOU MUST BE 18 YEARS OF AGE OR OLDER AND A FIRST-YEAR COLLEGE STUDENTS AT A PARTICIPATING UNIVERSITY. TO BE ELIGIBLE FOR CASH PRIZES TO BE AWARDED TO TOP SCORERS, YOU MUST PROVIDE YOUR UNIVERSITY-ISSUED EMAIL ADDRESS IN ORDER TO VERIFY YOUR ENROLLMENT AT A PARTICIPATING UNIVERSITY.

## How to Play

EACH WEEK BEGINS WITH A "QUESTION PERIOD" DURING WHICH YOU WILL ANSWER THE THREE CAMPUSGANDR QUESTIONS OF THE WEEK. EACH QUESTION WILL CONSIST OF TWO PARTS: ONE IN WHICH YOU WILL ATTEMPT TO GUESS HOW CLASSMATES WILL RESPOND AND ANOTHER WHERE YOU WILL REPORT YOUR OWN BEHAVIOR. AFTER ANSWERING THE THREE QUESTIONS, YOU WILL PLACE BETS ON THE ACCURACY OF YOUR GUESSES ABOUT CLASSMATES. NEXT YOU WILL HAVE THE OPTION OF PROGRESSING THROUGH THREE ADDITIONAL BRIEF PHASES OF PLAY: SIZE-UP, VOTING, AND SUBMISSION, WHICH OFFER OPPORTUNITIES TO SCORE ADDITIONAL POINTS. FIRST, DURING SIZE-UP, YOU WILL BE PRESENTED AT RANDOM WITH 3-4 BEHAVIORS REPORTED BY SAME AND OPPOSITE STUDENTS AT YOUR SCHOOL IN RESPONSE TO EACH OF THE 3 QUESTIONS OF THE WEEK AND ASKED TO "SIZE-UP" A HYPOTHETICAL CLASSMATE WHO SELECTED EACH RESPONSE ON 2 SLIDING SCALES FROM "TOGETHER" TO "HOT MESS" AND FROM "ATTRACTIVE" TO "UNATTRACTIVE". SECOND, DURING VOTING, HELP SELECT THE GANDR QUESTIONS FOR THE NEXT ROUND BY VIEWING POTENTIAL QUESTIONS SUBMITTED BY YOUR CLASSMATES AND DECIDING WHETHER TO "UPVOTE" OR "DOWNVOTE" EACH. FINALLY, DURING SUBMIT, YOU WILL HAVE THE OPPORTUNITY TO SUBMIT QUESTIONS OF YOUR OWN TO BE VOTED ON BY CLASSMATES. YOU WILL EARN POINTS FOR EVERY "SIZE-UP" YOU SUBMIT AND EVERY "VOTE" YOU CAST. ALSO, IF YOU SUBMIT A WINNING CAMPUSGANDR QUESTION (ONE THAT IS FEATURED IN A SUBSEQUENT ROUND) YOU WILL EARN SIGNIFICANT BONUS POINTS.

YOU WILL RECEIVE A NOTIFICATION AT THE END OF THE WEEK WHEN YOUR RESULTS ARE READY TO VIEW. TAPPING THIS NOTIFICATION WILL OPEN THE SCORING SELECTION SCREEN WHERE A SPINNER WILL SELECT TWO OF THE THREE WEEKLY QUESTIONS ON WHICH YOU WILL RECEIVE DETAILED FEEDBACK AND BE SCORED. NEXT, AN ANIMATED "RESULTS LOADING" SCREEN WILL DISPLAY PROFILE PHOTOS FOR ALL STUDENTS WHO ANSWERED THE CAMPUSGANDR QUESTIONS THAT WEEK AT YOUR SCHOOL.

DETAILED RESULTS WILL REVEAL HOW ACCURATE YOUR GUESSES ABOUT CLASSMATES WERE, THE POINTS YOU WON AND LOST, HOW YOUR BEHAVIORS COMPARE TO OTHER STUDENTS AT YOUR SCHOOL, AS WELL AS HOW "ATTRACTIVE" AND "TOGETHER" OTHER

### RISKS AND BENEFITS

You should be aware that Campusgandr questions of the week are user-generated and may ask about private, sensitive, or even "illegal" behaviors that could embarrass you or potentially get you in trouble (drinking, drug use, cheating) if your answers were shared with others. Rest assured that your secrets are safe with us (see the privacy policy that follows) and your individual responses to questions will NOT be shared with other users, administrators at your university, nor law enforcement officials. In addition, if you feel uncomfortable answering the questions, you can elect to skip specific questions or weeks of play entirely without penalty. You should be aware that you may find the detailed results you receive distressing. For example, it may be a real downer to learn that other students are studying much more than you or that other students rated the amount of partying you reported to be "unattractive" or a "hot mess". You may elect to quit playing campusgandr at any time.

CAMPUSGANDR IS INTENDED TO REDUCE UNCERTAINTY DURING THE TRANSITION TO COLLEGE OFFERING NEW COLLEGE STUDENTS HELPFUL AND ENTERTAINING SOCIAL INFORMATION ABOUT THEIR CLASSMATES AND NEW CAMPUS. IN ADDITION TO SOCIAL KNOWLEDGE, CAMPUSGANDR MAY ALSO OFFER YOU TO AN OPPORTUNITY TO WIN ONE OF SEVERAL SIZABLE CASH PRIZES (\$500, \$250, \$100) TO BE RAFFLED AT THE END OF THE SEMESTER. FOR EACH ROUND OF CAMPUSGANDR YOU PLAY, YOU WILL EARN AN ADDITIONAL ENTRY IN THE PRIZE RAFFLE. THUS, YOU CAN INCREASE YOUR CHANCES OF WINNING A PRIZE BY PLAYING MORE ROUNDS.

## GROUNDS FOR DISQUALIFICATION AND TERMINATION OF SERVICE

WE RESERVE THE RIGHT TO TERMINATE USE AND DISQUALIFY ANY USER FROM THE COMPETITION AT THEIR UNIVERSITY. GROUNDS FOR DISQUALIFICATION/TERMINATION INCLUDE BUT ARE NOT LIMITED TO ATTEMPTING TO CHEAT IN ANYWAY AND SUBMITTING QUESTIONS THAT MAY BE CONSIDERED OFFENSIVE TO OTHER USERS.

## DATA USAGE

IF YOU'RE USING THE APP OUTSIDE OF AN AREA WITH WI-FI, YOU SHOULD REMEMBER THAT YOUR TERMS OF AGREEMENT WITH YOUR MOBILE NETWORK PROVIDER WILL STILL APPLY. AS A RESULT, YOU MAY BE CHARGED BY YOUR MOBILE PROVIDER FOR THE COST OF DATA FOR THE DURATION OF THE CONNECTION WHILE ACCESSING THE APP, OR OTHER THIRD PARTY CHARGES. IN USING THE APP, YOU'RE ACCEPTING RESPONSIBILITY FOR ANY SUCH CHARGES, INCLUDING ROAMING DATA CHARGES IF YOU USE THE APP OUTSIDE OF YOUR HOME TERRITORY (I.E. REGION OR COUNTRY) WITHOUT TURNING OFF DATA ROAMING. IF YOU ARE NOT THE BILL PAYER FOR THE DEVICE ON WHICH YOU'RE USING THE APP, PLEASE BE AWARE THAT WE ASSUME THAT YOU HAVE RECEIVED PERMISSION FROM THE BILL PAYER FOR USING THE APP.

## APPLICATION UPDATES

THE CAMPUSGANDR TEAM IS COMMITTED TO ENSURING THAT THE APP IS AS USEFUL AND EFFICIENT AS POSSIBLE. FOR THAT REASON, WE RESERVE THE RIGHT TO MAKE CHANGES TO THE APP AT ANY TIME AND FOR ANY REASON. AT SOME POINT WE MAY WISH TO UPDATE THE APP. THE APP IS CURRENTLY AVAILABLE ON ANDROID AND IOS — THE REQUIREMENTS FOR BOTH SYSTEMS (AND FOR ANY ADDITIONAL SYSTEMS WE DECIDE TO EXTEND THE AVAILABILITY OF THE APP TO) MAY CHANGE, AND YOU'LL NEED TO DOWNLOAD THE UPDATES IF YOU WANT TO KEEP USING THE APP. WE CANNOT PROMISE THAT UPDATES ALWAYS WILL REMAIN RELEVANT TO YOU AND/OR WORK WITH THE IOS/ANDROID VERSION THAT YOU HAVE INSTALLED ON YOUR DEVICE. HOWEVER, YOU PROMISE TO ALWAYS ACCEPT UPDATES TO THE APPLICATION WHEN OFFERED TO YOU, WE MAY ALSO WISH TO STOP PROVIDING THE APP, AND MAY TERMINATE USE OF IT AT ANY TIME WITHOUT GIVING NOTICE OF TERMINATION TO YOU. UNLESS WE TELL YOU OTHERWISE, UPON ANY TERMINATION, (A) THE RIGHTS AND LICENSES GRANTED TO YOU IN THESE TERMS WILL END; (B) YOU MUST STOP USING THE APP, AND (IF NEEDED) DELETE IT FROM YOUR DEVICE.

## PRIVACY POLICY

LAST UPDATED 8 AUGUST 2018

CAMPUSGANDR ("WE" OR "US" OR "OUR") RESPECTS THE PRIVACY OF OUR USERS ("USER" OR "YOU"). THIS PRIVACY POLICY EXPLAINS HOW WE COLLECT, USE, DISCLOSE, AND SAFEGUARD YOUR INFORMATION WHEN YOU VISIT OUR MOBILE APPLICATION (THE "APPLICATION"). PLEASE READ THIS PRIVACY POLICY CAREFULLY. IF YOU DO NOT AGREE WITH THE TERMS OF THIS PRIVACY POLICY, PLEASE DO NOT ACCESS THE CAMPUSGANDR APPLICATION.

WE RESERVE THE RIGHT TO MAKE CHANGES TO THIS PRIVACY POLICY AT ANY TIME AND FOR ANY REASON. WE WILL ALERT YOU ABOUT ANY CHANGES BY UPDATING THE "LAST UPDATED" DATE OF THIS PRIVACY POLICY. YOU ARE ENCOURAGED TO PERIODICALLY REVIEW THIS PRIVACY POLICY TO STAY INFORMED OF UPDATES. YOU WILL BE DEEMED TO HAVE BEEN MADE AWARE OF, WILL BE SUBJECT TO, AND WILL BE DEEMED TO HAVE ACCEPTED THE CHANGES IN ANY REVISED PRIVACY POLICY BY YOUR CONTINUED USE OF THE APPLICATION AFTER THE DATE SUCH REVISED PRIVACY POLICY IS POSTED.

THIS PRIVACY POLICY DOES NOT APPLY TO THE THIRD-PARTY ONLINE/MOBILE STORE FROM WHICH YOU INSTALL THE APPLICATION. WE ARE NOT RESPONSIBLE FOR ANY OF THE DATA COLLECTED BY ANY SUCH THIRD PARTY.

## COLLECTION OF YOUR INFORMATION

WE MAY COLLECT INFORMATION ABOUT YOU IN A VARIETY OF WAYS. MUCH OF THE INFORMATION COLLECTED VIA THE APPLICATION DEPENDS ON YOUR ACTIONS AND THE PERMISSIONS YOU GRANT OR DENY WITHIN THE APPLICATION.

## PERSONAL DATA

INCLUDES DEMOGRAPHIC AND OTHER PERSONALLY IDENTIFIABLE INFORMATION THAT YOU VOLUNTARILY GIVE TO US WHEN ELECTING TO CREATE AN ACCOUNT TO PLAY IN CAMPUSGANDR. THIS DATA INCLUDES YOUR AGE IN YEARS, GENDER, AND UNIVERSITY ISSUED EMAIL ADDRESS, WHICH THE APPLICATION USES TO VERIFY THAT YOU ARE ENROLLED AT A PARTICULAR UNIVERSITY. THE APPLICATION ALSO EMPLOYS STANDARD SOCIAL MEDIA AUTHENTICATION OPTIONS FOR USER LOGIN AND COLLECTS LIMITED INFORMATION FROM YOUR SOCIAL MEDIA ACCOUNT IF YOU CHOOSE TO AUTHENTICATE VIA A SOCIAL MEDIA ACCOUNT AND GRANT CAMPUSGANDR THESE PERMISSIONS. DATA-RELATED INFORMATION ABOUT YOUR CAMPUSGANDR ACCOUNT AND SOCIAL MEDIA AUTHENTICATION ARE DETAILED IN THE NEXT SECTION.

## ACCOUNT DATA, SOCIAL MEDIA PERMISSIONS, & PRIVACY SETTINGS

YOU HAVE THE OPTION TO AUTHENTICATE WITH AN EXISTING SOCIAL MEDIA ACCOUNT (FACEBOOK/INSTAGRAM/TWITTER/SNAPCHAT) OR CREATING A NEW USERNAME AND PASSWORD AS WELL AS UPLOADING A PROFILE PHOTO MANUALLY. IF YOU CHOOSE TO AUTHENTICATE WITH SOCIAL MEDIA, YOU WILL BE PROMPTED TO ENTER YOUR CREDENTIALS FOR THE PLATFORM OF YOUR CHOICE AND THEN PERMIT OR DENY CAMPUSGANDR ACCESS TO YOUR YOUR EMAIL ADDRESS AND PROFILE PICTURE ASSOCIATED WITH THIS SOCIAL MEDIA ACCOUNT. THIS ALLOWS YOU TO SKIP THE STEPS ASSOCIATED WITH REGISTERING A NEW USERNAME A PASSWORD AND UPLOADING A PROFILE PHOTO. REGARDLESS OF WHETHER YOU CHOOSE TO CREATE YOUR ACCOUNT MANUALLY OR LOGIN WITH SOCIAL MEDIA CREDENTIALS, YOU WILL HAVE AN OPPORTUNITY TO COMPLETE A PUBLIC PROFILE WHICH INCLUDES ONLY YOUR PROFILE PHOTO (IF YOU CHOOSE TO PROVIDE ONE) COLLEGE MAJOR, HOMETOWN, AND A BRIEF BIO IN WHICH YOU CAN TELL OTHER PLAYERS A BIT ABOUT YOURSELF (SIMILAR TO AN INSTAGRAM OR TWITTER BIO). IF YOU CHOOSE TO CREATE A PUBLIC PROFILE IT WILL BE VIEWABLE TO OTHER USERS IN THE "PLAYERS" AREA OF THE APP. IMPORTANTLY, WITH THE EXCEPTION OF A 50X50 PIXEL THUMBNAIL VERSION OF YOUR PROFILE PHOTO, WHICH WILL BE INCLUDED IN A COLLAGE OF THE USERS AT YOUR UNIVERSITY WHO PLAY EACH WEEK IF YOU ALLOW IT TO BE, AND THIS OPTIONAL PUBLIC PROFILE THAT INCLUDES YOUR HOMETOWN, MAJOR, AND A BRIEF BIO IF YOU CHOOSE TO PROVIDE ONE, NONE OF YOUR PERSONAL DATA WILL BE VIEWABLE BY OTHER USERS ACCESSING THE APPLICATION. YOU CAN USE THE TOGGLE BUTTON IN APPLICATION SETTINGS TO ELECT TO, OR NOT TO, BE REPRESENTED BY YOUR PHOTO IN THE COLLAGE OF USERS PLAYING EACH ROUND AT YOUR UNIVERSITY. CAMPUSGANDR ALSO FEATURES A LEADERBOARD WHICH UPDATES FOLLOWING EACH ROUND OF PLAY TO DISPLAY USERS' PROFILE PHOTOS AND THEIR SCORES FROM HIGHEST TO LOWEST POINT TOTALS. YOU CAN USE TOGGLE BUTTONS IN THE APPLICATION SETTINGS TO INDICATE WHETHER OR NOT YOU WOULD LIKE TO BE VISIBLE TO OTHER STUDENTS AT YOUR SCHOOL IN THE IN THE LEADERBOARD AND/OR PUBLIC PROFILE AREA OF THE APP.

## DERIVATIVE DATA

INCLUDES INFORMATION OUR SERVERS AUTOMATICALLY COLLECT WHEN YOU ACCESS THE APPLICATION, SUCH AS YOUR NATIVE ACTIONS THAT ARE INTEGRAL TO THE APPLICATION, INCLUDING RESPONSES TO QUESTIONS OF THE WEEK, POINTS WAGERED, JUDGMENTS OF OTHER STUDENTS' BEHAVIORS, SUBMITTED QUESTIONS, QUESTION VOTES, AND POINTS SCORED, IMPORTANTLY NONE OF YOUR ACTIONS IN THE APP, INCLUDING YOUR ANSWERS TO QUESTIONS, WILL BE VIEWABLE BY OTHER USERS ACCESSING THE APPLICATION. IN APPLICATION SETTINGS YOU CAN, HOWEVER, CHOSE WHETHER, TO SHARE YOUR TOTAL SCORE WITH OTHER USERS BY HAVING IT INCLUDED WITH YOUR PROFILE PHOTO IN A LEADERBOARD WITHIN THE APPLICATION.

## MOBILE DEVICE DATA

DEVICE INFORMATION SUCH AS YOUR MOBILE DEVICE ID NUMBER, MODEL, MANUFACTURER, VERSION OF YOUR OPERATING MAY BE LOGGED BY OUR SERVER.

## **PUSH NOTIFICATIONS**

WE WILL REQUEST TO SEND YOU PUSH NOTIFICATIONS REGARDING YOUR ACCOUNT OR THE APPLICATION. PUSH NOTIFICATIONS MAY ALERT YOU TO NEW ROUNDS OF PLAY OPENING, NEW RESULTS BEING AVAILABLE FOR YOU TO VIEW, THE LEADERBOARD BEING UPDATED, A QUESTION YOU SUBMITTED BEING FEATURED AS A QUESTION OF THE WEEK AT YOUR SCHOOL, ETC. IF YOU WISH TO OPT-OUT FROM RECEIVING THESE TYPES OF COMMUNICATIONS, YOU MAY TURN THEM OFF IN YOUR DEVICE'S SETTINGS.

## **USE OF YOUR INFORMATION**

HAVING ACCURATE INFORMATION ABOUT YOU PERMITS US TO PROVIDE YOU WITH A SMOOTH, EFFICIENT, AND CUSTOMIZED EXPERIENCE. SPECIFICALLY, WE MAY USE INFORMATION COLLECTED ABOUT YOU VIA THE APPLICATION TO:

- NOTIFY YOU IN THE EVENT YOU WIN A CASH PRIZE AS A TOP SCORER AT YOUR UNIVERSITY.
- COMPILE ANONYMOUS STATISTICAL DATA AND ANALYSIS FOR INTERNAL USE.
- CREATE AND MANAGE YOUR ACCOUNT.
- 4. ALLOW YOU TO VIEW THE OTHER STUDENTS PLAYING AT YOUR UNIVERSITY.
- ALLOW YOU TO SEE HOW ACCURATELY YOU VIEW THE BEHAVIORS AND ATTITUDES OF CLASSMATES
- 6. ALLOW YOU TO SEE HOW YOUR BEHAVIORS AND ATTITUDES COMPARE TO, AND ARE JUDGED BY CLASSMATES.
- 7. CALCULATE THE POINTS YOU WIN AND LOSE EACH ROUND AND TRACK YOUR SCORE ACROSS ROUNDS OF PLAY.
- 8. GENERATE A PERSONAL PROFILE TO MAKE YOUR FUTURE VISITS TO THE APPLICATION MORE PERSONALIZED.
- 9. INCREASE THE EFFICIENCY AND OPERATION OF THE APPLICATION. MONITOR AND ANALYZE USAGE AND TRENDS TO IMPROVE YOUR EXPERIENCE WITH THE APPLICATION.
- 11. NOTIFY YOU OF UPDATES TO THE APPLICATION.
- 12. REQUEST FEEDBACK AND CONTACT YOU ABOUT YOUR USE OF THE APPLICATION.
- 13. RESOLVE DISPUTES AND TROUBLESHOOT PROBLEMS.
- 14. RESPOND TO PRODUCT AND CUSTOMER SERVICE REQUESTS.
- 15. SEND YOU A NEWSLETTER.

## DISCLOSURE OF YOUR INFORMATION

CAMPUSGANDR WILL NOT SHARE YOUR PERSONAL, FACEBOOK, DERIVATIVE, OR MOBILE DEVICE DATA WITH THIRD PARTIES.

## TRACKING TECHNOLOGIES

#### WEBSITE ANALYTICS

WE MAY ALSO PARTNER WITH SELECTED THIRD-PARTY ANALYTICS VENDORS SUCH AS ADOBE ANALYTICS, GOOGLE ANALYTICS, AND/OR HEAP ANALYTICS TO ALLOW TRACKING TECHNOLOGIES ON THE APPLICATION THROUGH THE USE OF FIRST PARTY COOKIES AND THIRD-PARTY COOKIES, TO, AMONG OTHER THINGS, ANALYZE AND TRACK USERS' USE OF THE APPLICATION, DETERMINE THE POPULARITY OF CERTAIN CONTENT, AND BETTER UNDERSTAND APPLICATION USAGE. BY ACCESSING THE APPLICATION, YOU CONSENT TO THE COLLECTION AND USE OF YOUR INFORMATION BY THESE THIRD-PARTY VENDORS. YOU ARE ENCOURAGED TO REVIEW THEIR PRIVACY POLICY AND CONTACT THEM DIRECTLY FOR RESPONSES TO YOUR QUESTIONS. WE DO NOT TRANSFER PERSONAL INFORMATION TO THESE THIRD-PARTY VENDORS.

## SECURITY OF YOUR INFORMATION

WE EMPLOY THE MOST ADVANCED TECHNOLOGIES AND INTERNAL PROTOCOLS (LAYERED SECURITY, HTTPS PROTOCOL, SSL CERTIFICATES, TSL ENCRYPTION IN TRANSIT, ETC.) TO TRANSMIT, SECURE, AND STORE AND PROTECT ALL APPLICATION DATA. THESE PROTOCOLS SAFEGUARD PRIVACY BETWEEN COMMUNICATING APPLICATIONS AND THEIR USERS ON THE INTERNET. ALSO USED TO SECURE BANK AND CREDIT CARD TRANSACTIONS ONLINE, THESE PROTOCOLS ENSURE THAT NO THIRD PARTY MAY EAVESDROP OR TAMPER WITH SUBMITTED DATA.

## POLICY FOR CHILDREN

WE DO NOT KNOWINGLY SOLICIT INFORMATION FROM OR MARKET TO CHILDREN UNDER THE AGE OF 18. IF YOU BECOME AWARE OF ANY DATA WE HAVE COLLECTED FROM CHILDREN UNDER AGE 18, PLEASE CONTACT US USING THE CONTACT INFORMATION PROVIDED BELOW.

## CONTROLS FOR DO-NOT-TRACK FEATURES

MOST WEB BROWSERS AND SOME MOBILE OPERATING SYSTEMS [AND OUR MOBILE APPLICATIONS] INCLUDE A DO-NOT-TRACK ("DNT") FEATURE OR SETTING YOU CAN ACTIVATE TO SIGNAL YOUR PRIVACY PREFERENCE NOT TO HAVE DATA ABOUT YOUR ONLINE BROWSING ACTIVITIES MONITORED AND COLLECTED. NO UNIFORM TECHNOLOGY STANDARD FOR RECOGNIZING AND IMPLEMENTING DNT SIGNALS HAS BEEN FINALIZED. AS SUCH, WE DO NOT CURRENTLY RESPOND TO DNT BROWSER SIGNALS OR ANY OTHER MECHANISM THAT AUTOMATICALLY COMMUNICATES YOUR CHOICE NOT TO BE TRACKED ONLINE. IF A STANDARD FOR ONLINE TRACKING IS ADOPTED THAT WE MUST FOLLOW IN THE FUTURE, WE WILL INFORM YOU ABOUT THAT PRACTICE IN A REVISED VERSION OF THIS PRIVACY POLICY.

## OPTIONS REGARDING YOUR INFORMATION

**ACCOUNT INFORMATION** 

YOU MAY AT ANY TIME REVIEW OR CHANGE THE INFORMATION IN YOUR ACCOUNT OR TERMINATE YOUR ACCOUNT BY:

- LOGGING INTO YOUR ACCOUNT SETTINGS AND UPDATING YOUR ACCOUNT
- CONTACTING US USING THE CONTACT INFORMATION PROVIDED BELOW

UPON YOUR REQUEST TO TERMINATE YOUR ACCOUNT, WE WILL DEACTIVATE OR DELETE YOUR ACCOUNT AND INFORMATION FROM OUR ACTIVE DATABASES. HOWEVER, SOME INFORMATION MAY BE RETAINED IN OUR FILES TO PREVENT FRAUD, TROUBLESHOOT PROBLEMS, ENFORCE OUR TERMS OF USE AND/OR COMPLY WITH LEGAL REQUIREMENTS.]

## **EMAILS AND NOTIFICATIONS**

IF YOU NO LONGER WISH TO RECEIVE EMAILS AND PUSH NOTIFICATIONS FROM US, YOU MAY OPT-OUT BY:

- Noting your preferences at the time you register your account with the Application
- LOGGING INTO YOUR ACCOUNT SETTINGS AND UPDATING YOUR PREFERENCES
- CONTACTING US USING THE CONTACT INFORMATION PROVIDED BELOW

## CALIFORNIA PRIVACY RIGHTS

CALIFORNIA CIVIL CODE SECTION 1798.83, ALSO KNOWN AS THE "SHINE THE LIGHT" LAW, PERMITS OUR USERS WHO ARE CALIFORNIA RESIDENTS TO REQUEST AND OBTAIN FROM US, ONCE A YEAR AND FREE OF CHARGE, INFORMATION ABOUT CATEGORIES OF PERSONAL INFORMATION (IF ANY) WE DISCLOSED TO THIRD PARTIES FOR DIRECT MARKETING PURPOSES AND THE NAMES AND ADDRESSES OF ALL THIRD PARTIES WITH WHICH WE SHARED PERSONAL INFORMATION IN THE IMMEDIATELY PRECEDING CALENDAR YEAR. IF YOU ARE A CALIFORNIA RESIDENT AND WOULD LIKE TO MAKE SUCH A REQUEST, PLEASE SUBMIT YOUR REQUEST IN WRITING TO US USING THE CONTACT INFORMATION PROVIDED BELOW.

## **CONTACT US**

IF YOU HAVE QUESTIONS OR COMMENTS ABOUT CAMPUSGANDR'S DATA PRIVACY, TERMS OR CONDITIONS PLEASE CONTACT THE CAMPUSGANDR TEAM AT:

[310-568-8661] [INFO@CAMPUSGANDR.COM]

## Informed Consent Form- CampusGANDR Evaluation Study (RCT)

You are invited to participate in a research project being conducted by the researchers in the Psychology Department at [Loyola Marymount University/ University of Houston]. This informed consent form describes the study and tells you what you can expect if you become a participant. Please read it carefully before checking one of the boxes at the end.

#### **ELIGIBILITY**

As a registered first-year [LMU/UH] student at playing CampusGANDR, you are invited to participate in a special study designed to evaluate the app. To participate in this study you must be between 18 and 20 years old and be willing to play the game weekly during the Fall semester, and complete three surveys over the next year.

#### **PURPOSE**

As you know, CampusGANDR is a new app which invites first-year college students to test their social percptions, learn about classmates, and discover truths about life on campus all while having an opportunity to win cash prizes of ranging from \$100 to \$500. Each week during the fall semester, guess about classmates' attitudes and behaviors and then wager poins on the accuracy of each guess. Win wagered points for accurate guesses and lose wagered points for inaccurate guesses. This study is being conducted to test the CampusGANDR app at two universities and improve it before it is released to the public. Playing CampusGANDR will take no more than 5-6 minutes per week and the 4 surveys you will complete in this study will each take no longer than 20 minutes to complete. Survey questions will ask you about your preferences for smartphone applications and include questions about your academic and social life at LMU.

#### **DATA USE**

While CampusGANDR is meant to be entertaining, it also designed to be a valuable tool for reducing uncertainty during the transition to college, learning about new classmates, acclimating you to life on campus. As such, your responses to survey questions may be aggregated with data collected within the app and, along with the responses of other users, be used in the research programs of CampusGANDR project personnel affiliated with [UH/LMU]. All research reports will focus on highlighting group trends rather than individual responses. A description of this clinical trial will be available on http://www.ClinicalTrials.gov. This website will not include information that can identify you as a participant in this research. At most, the website will include a summary of the results. You can search this website at any time.

#### **CONFIDENTALITY & DATA SECURITY**

When you registered for CampusGANDR, you provided information for a brief user profile and were given the option of permitting CampusGANDR to use a profile photo from one of your social media accounts, uploading another photo to represent you in the app, or remaining faceless. It is important to understand that NONE of your social media account or CampusGANDR profile information will be linked to your responses to evaluation study survey questions. You were also given the option of having your profile picture and total round scores posted in a leaderboard visible to other authenticated CampusGANDR players in your class. These privacy options can be changed at any time in the Settings sections of the app. Whether you provide a profile photo or opt to make yourself visible in the leaderboard is entirely up to you, and not required to play CampusGANDR or participate in this evaluation study. It is important to understand that if you choose to provide a profile photo and/or be included in the leaderboard, you may be recognized by your classmates as a CampusGANDR player, and also recognize these classmates as CampusGANDR players. However, the other students playing CampusGANDR at your school will NOT know that you participating in this evaluation study unless you personally disclose this information to them. Your participation in this evaluation study is strictly confidential which means that you will not be identified as a participant in this study and the research team will not link your responses to survey items or CampusGANDR questions to your name or contact information. For this purpose, there will be an arbitrarily assigned sequence number on all your questionnaires and study data. The purpose of this sequence number is to keep track of materials collected in the study to be used in data analyses. Information regarding your first name, contact information, participant ID number, and whether or not each aspect of the study has been completed will be kept separate from the actual data at all times. This will

ensure that the data provided from the study will always be associated with a participant ID number and will never be connected directly with any names or identifying information. These will be locked in cabinets accessible to the Principal Investigators and research staff only. Moreover, examination of the study data will focus on highlighting group trends and not individual responses.

To help keep your information confidential, the current project has a Confidentiality Certificate from the U.S. Department of Health and Human Services (DHHS). This protects the investigators from being forced, even under a court order or subpoena, to release information that could identify you. Please be aware, however, that if harm to you or others becomes a concern, the researchers may choose to provide information to appropriate individuals or agencies. For example, should such a situation arise, the research team may contact Student Psychological Services. Also, because this research is sponsored by the National Institute of Alcoholism and Alcohol Abuse, staff from that institute may review records that identify you only for audit or program evaluation purposes. Despite the presence of the Certificate of Confidentiality, you are responsible for actively maintaining your confidentiality as a participant in this project. A Confidentiality Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research. All data transmitted within CampusGANDR app and the online surveys you will complete as a participant in this study is protected by Transport Layer Security (TLS) encryption (also known as HTTPS), which is a protocol that ensures privacy between communicating applications and their users on the Internet. Also used to secure bank and credit card transactions online, TLS ensures that no third party may eavesdrop or tamper with submitted data.

#### **POTENTIAL RISKS & BENEFITS**

CampusGANDR questions of the week are user-generated and may ask about private, sensitive, or even "illegal" behaviors that could embarrass you or potentially get you in trouble (drinking, drug use, cheating) if your answers were shared with others. Similarly, questions in this survey study may also ask about sensitive or private health-related topics related to the transition to college (i.e., alcohol use, drug use, depression, anxiety, stress). Rest assured that the answers you provide will NOT be shared with other CampusGANDR users, study participants, administrators at your university, nor law enforcement officials. In addition, if you feel uncomfortable answering the questions, you can elect to skip specific questions or weeks of play entirely without penalty. You may elect to quit playing CampusGANDR at any time and/or choose withdrawal from this study at any time. Campusgandr is intended to reduce uncertainty during the transition to college by offering new college students helpful and entertaining social information about their classmates and new campus. Learning what other students find attractive as well as how much time other students really spend studying, engaging in service, socializing, and partying may quell your curiosities and provide special insight that may help you prioritize your busy life on campus. Your participation in this evaluation study will help shape the app for future cohorts of first-year students.

#### **INCENTIVES**

Participants who complete the first survey and play the first CampusGANDR round will receive an email within one business day containing an e-gift card for \$20. The three follow-up surveys will be of similar length and will also include a \$20 gift card. In addition, students who successfully complete all four surveys will receive an additional \$20 bonus after the final survey, for a total of \$100 from the surveys. You will also earn incentives for simply playing CampusGANDR each week. Every four weeks during the Fall semester gift cards for \$10 will be sent to all students who played at least 3 of the 4 intervening GANDR rounds. Play will last for a total of 12 weeks, resulting in \$30 worth of incentives for CampusGANDR play. Thus, direct incentives total \$130. In addition to these incentives for study participation, all students playing CampusGANDR at [LMU/UH] will be eligible for winning cash prizes awarded to the top scorers at each University each month over the Fall semester. As a participant in this evaluation study you remain eligible for these top scorer cash prizes.

#### FOR MORE INFORMATION

Dr. [Joe LaBrie/Clayton Neighbors] can be reached at [address], office phone number [phone number], [email address], if you have any questions or concerns about your participation in CampusGANDR.

If you have questions regarding your rights as a research subject, you may contact Dr. [IRB Chair], Chair of the Human Subjects Review Committee, at [phone], [email].

| | By checking this box, I acknowledge that: • I would like to play CampusGANDR and participate in this evaluation study. |
|---|---|
| | By checking this box, I acknowledge that: • I do not wish to participate in this evaluation study and/or CampusGANDR |
| I, | , affirm that I have read and understood the above statement and |
| have I | nad all of my questions answered. |
| Date: | |
| Electr | onic Signature: |

Please check ONE of the boxes below: